CLINICAL TRIAL: NCT02749929
Title: A Double-blind Placebo-controlled Study of Low-level Laser Therapy in Wrist Fractures
Brief Title: Low-level Laser Therapy in Wrist Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Principal Investigator, Humaira Sæbø, MS, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 569093
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Colles' Fracture
Keywords: Distal radius fracture, Low Level Laser Therapy
MeSH Terms: conditions — Colles' Fracture; Wrist Fractures | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Level Laser therapy (Experimental): After inclusion in the study, a small window of approximately 1 cm2 opening will be made in the cast in order for the laser to make skin contact. The laser is a super pulsed infrared laser with a wavelength of 904 nm, belonging to laser class 3B. The light from the laser is not visible to the eye, and will not give any perceptible stimulus.
  Low-Level Laser therapy (LLLT) will be given according to the recommended dosage from World Association of Laser Therapy (WALT). A LLLT dose of 3.6 Joules will be administered at two points over the fracture site.
  Interventions: Other: Low level laser therapy
- Placebo Low-Level Laser therapy (Placebo Comparator): After inclusion in the study, a small window of approximately 1 cm2 opening will be made in the cast in order for the placebo laser to make skin contact. The placebo laser is identical in apperance to a super pulsed infrared laser with a wavelength of 904 nm, belonging to laser class 3B. Since the light from the laser is invisible, neither the participant nor the therapist will know whether the laser is a placebo. The treatment time and number of treated points will be identical to group 1.
  Interventions: Other: Placebo Low Level Laser Therapy

INTERVENTIONS:
Other: Low level laser therapy — The laser is an infrared (invisible) 60 mW 904 nm Irradia Midlaser
  Arms: Low-Level Laser therapy
Other: Placebo Low Level Laser Therapy — The placebo laser is an identical device to the active laser, made by Irradia Midlaser
  Arms: Placebo Low-Level Laser therapy

SUMMARY:
Approximately 15,000 persons in Norway suffer from wrist fractures during a year, making it the most prevalent fracture in this country. Treated conservatively, a cast is used for 4-6 weeks before removal. After discontinuation of the cast, physiotherapy is implemented to aid in improving range of motion and regaining function of the injured wrist. The pain after injury can affect the patient to a greater or lesser extent, and it is common to prescribe sick leave for shorter amounts of time after the injury.

Studies suggest that a physiotherapy intervention with Low Level Laser therapy (LLLT) may reduce pain and swelling after acute trauma, and potentially promote healing. The aim of this study is to evaluate the effect of LLLT on pain and function at 2, 4, 8 and 26 weeks after injury.

DETAILED DESCRIPTION:
Patients with wrist fractures are recruited from Bergen Municipal Emergency Ward, where they are randomly divided into two groups with concealed allocation. The fracture is immobilized with a cast, with a small opening where Low Level Laser therapy can be administered in skin contact. The patients will receive treatment 3 times a week, for 3 weeks. After discontinuation of the cast, the patients swelling, pain, grip strength and function of the wrist is measured. The patients will meet for follow-up controls until 26 weeks after injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal radiusfraktur, with or without ulna fracture Colles' fracture
* The breach must be closed
* Under 10 degrees dorsal displacement of radius
* Under 5mm shortening of the radius
* Under 3 mm step in the joint
* 18+ years

Exclusion Criteria:

* People who do not speak Norwegian or English
* If the patient is pregnant
* Patient with Smith fracture
* Wounds over fracture area
* If the patient have a peripheral nerve injury
* If the patient had (previously) operated wrist
* Persons with verified osteoporosis at the time of injury, systemic inflammatory disease (rheumatism), mental illness, stroke, Parkinson's disease, multiple sclerosis, cancer or congenital malformations in wrist
* If the laser treatment can not be started within 3 days after fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-04; Primary Completion 2020-11-30 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Function and pain | 26 weeks
  Function and will be assessed using Patient Rating Wrist and Hand Evaluation a (PRWHE), and questions about night pain/pain killers

SECONDARY OUTCOMES:
Pain by pressure | 26 weeks
  Pain Pressure Threshold over distal radius will be assessed using Pressure Algometry
Swelling | 26 weeks
  Swelling will be assessed using measurement tape
Active range of motion | 26 weeks
  Active range of motion will be assessed using goniometer
Grip- and pinch Strength | 26 weeks
  Strength will be assessed using handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Jan Magnus Bjordal, Professor, Study Director — University of Bergen
Locations (1):
- Bergen Accident Emergency Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No